CLINICAL TRIAL: NCT06080061
Title: Phase I Trial of Personalized Accelerated ChEmoRadiation (PACER) for Lung Cancer
Brief Title: Personalized Accelerated ChEmoRadiation (PACER) for Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: LUNGevity Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-71744; NCI-2024-00696 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hypofractionated accelerated radiation therapy (HART) (Experimental): Patients will either be treated with 60-66 Gy in 30, 25, or 20 fractions based on ability to meet constraints to key organs at risk
  Interventions: Radiation: Hypofractionated accelerated radiation therapy

INTERVENTIONS:
Radiation: Hypofractionated accelerated radiation therapy — Hypofractionated accelerated radiation therapy

SUMMARY:
The purpose of this study is to examine the use of hypofractionated accelerated radiation therapy (HART) to treat locally advanced lung cancer. Depending on the location and size of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented malignancy of the lung including non-small cell lung cancer or small cell lung cancer planned for definitive therapy with fractionated radiation (60-66 Gy) and concurrent systemic therapy
* ECOG performance status of 0-2
* Age > 18 years old
* Ability to understand and the willingness to personally sign the written IRB approved informed consent document
* Estimated life expectancy of 12 weeks or longer

Exclusion Criteria:

* Contraindication to receiving radiotherapy or systemic therapy as determined by treating radiation and medical oncologist
* Age < 18 years old
* Tumor directly invading the major pulmonary arteries, aorta, heart or proximal bronchial tree
* Diagnosis of interstitial pulmonary fibrosis
* Previous radiation therapy to the thorax that would result in overlapping high dose radiation fields

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting pulmonary and esophageal toxicity | 9 months
  Toxicities will be scored by the CTCAE v5.0 criteria. Specific toxicities evaluated are grade 2+ pneumonitis and grade 3+ esophagitis as well as other G3+ pulmonary, esophageal or cardiac toxicities that could be probably or definitely attributed to rT.

SECONDARY OUTCOMES:
Acute and Late Toxicities | 36 months
  Patients will be evaluated by the rates of acute and late grade 2+ toxicities including lung, esophageal, cardiac, chest wall, and neurologic.
Integrated adaptive dosing regimen with an automated planning system | 36 months
  Evaluating the feasibility of integrating an adaptive dosing regimen with an automated planning system with the percentage of automated plans used and the time to plan approval.
Progression free survival | 36 months
  Determine progression free survival in patients treated with hypofractionated radiation therapy with concurrent systemic therapy
Overall survival | 36 months
  Determine overall survival in patients treated with hypofractionated radiation therapy with concurrent systemic therapy
Local control | 36 months
  Determine local control in patients treated with hypofractionated radiation therapy with concurrent systemic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lucas K Vitzthum, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States